CLINICAL TRIAL: NCT03154944
Title: A Clinical Investigation Evaluating Three New 1-piece Ostomy Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CP275
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ostomy device 1 (Experimental): In this arm the subjects test a new ostomy device consisting of a known adhesive and a new top film
  Interventions: Device: Ostomy device 1
- Ostomy device 2 (Experimental): In this arm the subjects test a new ostomy device consisting of a new adhesive and a known top film
  Interventions: Device: Ostomy device 2
- Ostomy device 3 (Experimental): In this arm the subjects test a new ostomy device consisting of a known adhesive and a new top film
  Interventions: Device: Ostomy device 3

INTERVENTIONS:
Device: Ostomy device 1 — This device consists of a known adhesive and a new top film
  Arms: Ostomy device 1
Device: Ostomy device 2 — This device consists of a new adhesive and a known top film
  Arms: Ostomy device 2
Device: Ostomy device 3 — This device consists of a known adhesive and a new top film
  Arms: Ostomy device 3

SUMMARY:
This investigation evaluates three new ostomy appliances and their impact on the peristomal skin.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent and in DK: signed a letter of authority
2. Be at least 18 years of age and have full legal capacity
3. Have had their ileostomy for at least 3 months
4. Have an ileostomy with a diameter between 10 and 55 mm
5. Be able to handle the Clinical App. and product themselves
6. Must be able to use custom cut product
7. Minimum change of product every second day
8. If current product is SenSura Mio - Be willing to use Maxi bag during investigation
9. Subject using Sensura or Sensura Mio flat 1 pc. open for at least two weeks before inclusion in the study.
10. Negative result of a pregnancy test for women of childbearing age (only DK)

Exclusion Criteria:

1. Are currently receiving or have within the past 2 months received radio-and/or chemotherapy (low doses chemotherapy are allowed for other indications than cancer, e.g. below 15 mg methotrexate for rheumatoid arthritis)
2. Are currently receiving or have within the past month received topical steroid treatment in the peristomal skin area, e.g. lotion or spray. Systemic steroid treatment (e.g. injection, or tablet) are allowed.
3. Are pregnant or breastfeeding**
4. Are participating in other interventional clinical investigations or have previously participated in this investigation
5. Are currently suffering from peristomal skin problems i.e. bleeding and/or broken skin (assessed by the investigator)
6. Have known hypersensitivity towards any of the products used in the investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birte P Jakosen, MD, Principal Investigator — Medial director
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ostomy Device 1 | Ostomy Device 2 | Ostomy Device 3
Started | 13 | 15 | 10
Completed | 13 | 15 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ostomy Device 1 | Ostomy Device 2 | Ostomy Device 3 | Total
Number analyzed (Participants) | 13 | 15 | 10 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (6.4) | 70.1 (7.7) | 63.6 (13) | 68.4 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 11 | 13 | 7 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 13 | 15 | 10 | 38

OUTCOME MEASURES:

1. Primary Outcome: Trans Epidermal Water Loss
Description: The trans epidermal water loss is measured on the peristomal skin using a probe. The Tran epirdermal water loss is a maesure for the skins barrier function. There is always a loss of water from the skin due to natural evaporation. However, when the skin barrier is damaged the evaporation of water increases leading to a higher trans epidermal water loss. Thus, trans epidermal water loss is used to assess the damage to the skin. Measurements are in grams of water per square meter per hour (g/m^2/h).
Time Frame: 7 days
Measure: Least Squares Mean (95% Confidence Interval); unit: g/m^2/h
Arm/Group | Ostomy Device 1 | Ostomy Device 2 | Ostomy Device 3
Number analyzed (Participants) | 13 | 15 | 10
g/m^2/h | 19.6 [15.5 to 24.9] | 20.7 [16.6 to 25.8] | 24.1 [18.2 to 31.8]

ADVERSE EVENTS:
Time Frame: 42 days
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research
Arm/Group | Ostomy Device 1 | Ostomy Device 2 | Ostomy Device 3
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/15 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15 | 0/10
Other Adverse Events (participants affected / at risk) | 2/13 | 1/15 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ostomy Device 1 (N=13) | Ostomy Device 2 (N=15) | Ostomy Device 3 (N=10)
Peristomal skin complications (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (2) — Peristomal skin complications

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT03154944/Prot_SAP_000.pdf